CLINICAL TRIAL: NCT04562337
Title: SHR-1316 Plus Chemotherapy and Sequential Thoracic Radiotherapy as First-line Therapy for Extensive-stage Small-Cell Lung Cancer (ES-SCLC): a Phase II Trial
Brief Title: SHR-1316 Combined With Chemotherapy and Chest Radiotherapy in ES-SCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinming Yu, President of Shandong Cancer Hospital and Institute, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ES-SCLC-1st-IIT-SHR1316-CRT
Record Dates: First submitted 2020-08-28; First posted 2020-09-24 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Extensive-stage Small Cell Lung Cancer
Keywords: SHR1316, Chemotherapy, Radiotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Carboplatin; Etoposide; Radiotherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR1316+Chemotherapy +Radiotherapy (Experimental): Paiticipant receive SHR-1316 、Chemotherapy and Radiotherapy
  Interventions: Drug: SHR1316; Drug: Carboplatin; Drug: Etoposide; Radiation: Radiation therapy; Drug: Cisplatin

INTERVENTIONS:
Drug: SHR1316 — Anti-PD-L1 antibody
  Other Names: Adebrelimab
Drug: Carboplatin — Carboplatin intravenous infusion will be administered during the induction phase (Cycles 1-4 or 6).
Drug: Etoposide — Etoposide intravenous infusion will be administered during the induction phase (Cycles 1-4 or 6).
Radiation: Radiation therapy — Thoracic radiation therapy ,TRT
Drug: Cisplatin — Cisplatin intravenous infusion will be administered during the induction phase (Cycles 1-4 or 6).

SUMMARY:
This study is a one arm, open, single center phase II study. The main purpose of this study was to evaluate the tolerance and preliminary efficacy of SHR1316 combined with chest radiotherapy after induction therapy.

DETAILED DESCRIPTION:
This is a single-arm, single-center phase II study. Eligible subjects will receive the following treatment regimens: 4~6 cycles of SHR1316 combined with EP/EC (etoposide, 100mg/m2, D1-3, q3w and cisplatin, 75mg/m², D1, q3w or carboplatin, AUC=5, D1, q3w). Patients with response sequentially received adebrelimab combined with chest radiotherapy based on investigator decision. Patients then the maintenance therapy with adebrelimab until disease progression or intolerable AEs.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Extensive small cell lung cancer
* Eastern Cooperative Oncology Group performance status (PS) of 0 to 1
* 18 to 75 years old
* The function of vital organs meets the following requirements. WBC ≥ 3.0 × 10^9/L, ANC≥1.5×10^9/L, PLT≥100×10^9/L, Hb≥9g/dL, ALT and AST ≤2.5 times ULN, TBIL ≤1.5 x ULN, CREA ≤1.5 times ULN or CCr≥50mL/min. INR≤1.5 x ULN, APTT ≤1.5 x ULN
* have not received first-line systemic therapy or immunosuppressive therapy for es-sclc
* The estimated survival period is more than 8 weeks
* With measurable lesion defined by the RECIST v1.1: Previously irradiated lesions may only be considered as measurable disease if disease progression has been unequivocally documented at that site since radiation and the previously irradiated lesion is not the only site of disease;
* Signed written informed consent prior to study entry

Exclusion Criteria:

* Active or untreated CNS metastases
* Leptomeningeal diseases
* Uncontrolled or symptomatic hypercalcemia
* Active, known or suspected autoimmune diseases
* have received any T cell co stimulation or immune checkpoint therapy
* Corticosteroids (> 10 mg / day prednisone or equivalent) or other immunosuppressants were used within 14 days before the first dose of study drug.
* Subjects had active infections.
* Failing to properly control the clinical symptoms or disease of the heart
* Patients who have previously received allogeneic bone marrow transplantation or solid organ transplantation
* Known to be allergic to the study drug or excipients, known to have a serious allergic reaction to any kind of monoclonal antibody; have a history of hypersensitivity to cisplatin or etoposide
* According to the researcher's judgment, there are other factors that may lead to the termination of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
overall survival （OS） | Up to approximately 36 months

SECONDARY OUTCOMES:
progression-free survival (PFS) | Up to approximately 36 months
Objective Response Rate (ORR) | Up to approximately 36 months
disease control rate (DCR) | Up to approximately 36 months
Duration of Response (DOR) | Up to approximately 36 months
Adverse events | Up to approximately 36 months
  Safety, incidence and severity of adverse events (AEs) and serious adverse events (SAEs) per CTCAE 5.0 criteria
6- and 12-month PFS rates | 6 Months and 12 Months
  Percentage of Participants Alive and Without PD, as Assessed by the Investigator Using RECIST v1.1, at 6 Months and 12 Months
1- and 2-year OS rates | 1 Year and 2 Years
  Percentage of Participants Alive at 1 Year and 2 Years

OTHER OUTCOMES:
Change of ctDNA status | Up to approximately 36 months
  Change of circulating tumor DNA (ctDNA) status in blood before and after receving treatment

CONTACTS AND LOCATIONS:
Overall Officials: JinMing Yu, PhD, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen D, Zou B, Li B, Gao A, Huang W, Shao Q, Meng X, Zhang P, Tang X, Hu X, Zhang Y, Guo J, Zhao C, Yuan J, Li Q, Zhu C, Yu J, Wang L. Adebrelimab plus chemotherapy and sequential thoracic radiotherapy as first-line therapy for extensive-stage small-cell lung cancer (ES-SCLC): a phase II trial. EClinicalMedicine. 2024 Aug 21;75:102795. doi: 10.1016/j.eclinm.2024.102795. eCollection 2024 Sep. PMID 39252865